CLINICAL TRIAL: NCT04492072
Title: Misoprostol With Mechanical Dilation Versus Oxytocin With Mechanical Dilation for High-risk Pregnancy Inductions: A Randomized Control Trial
Brief Title: Misoprostol With Mechanical Dilation Versus Oxytocin With Mechanical Dilation for High-risk Pregnancy Inductions
Acronym: MODE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Leen Al-Hafez, Principal Investigator, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20D.435
Record Dates: First submitted 2020-07-17; First posted 2020-07-30 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Cesarean Section; Misoprostol; Oxytocin; High Risk Pregnancy
MeSH Terms: interventions — Oxytocin; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin with Mechanical Dilation (Experimental): If the patient is randomized to Cook Balloon and Oxytocin - The balloon inflated to 60cc will be placed and oxytocin 2 mu/min will be initiated, and increased incrementally by 2mu/min every 30 minutes. If the cook cannot be placed initially, it will be reattempted and placed within 6 hours of oxytocin starting. The Cook catheter will remain in place until spontaneously expelled, or if not, after 12 hours of placement.
  If a Cook Balloon is not available, a Foley catheter can be used in its place as alternate and equivalent form of mechanical dilation.
  Interventions: Drug: Oxytocin
- Misoprostol with Mechanical Dilation (Active Comparator): If the patient is randomized to Misoprostol and Cook balloon - she will be given 25mcg of misoprostol orally or buccal and a Cook Balloon inflated to 60cc will be placed. She will subsequently receive 50mcg oral or buccal misoprostol every 4 hours up to 4 doses. If regular contractions occur (three or more contractions in a 10-minute period), the patient will be switched to Oxytocin 2 mu/min, and increased incrementally by 2mu/min every 30 minutes. If the cook balloon cannot be placed initially, it will be reattempted and placed within 6 hours of induction start. The Cook catheter will remain in place until spontaneously expelled, or at the fourth misoprostol administration. At this point, oxytocin will be started if not already initiated and artificial rupture of membranes will occur
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Oxytocin — Intervention
  Other Names: Mechanical Dilation
  Arms: Oxytocin with Mechanical Dilation
Drug: Misoprostol — Control
  Other Names: Mechanical Dilation
  Arms: Misoprostol with Mechanical Dilation

SUMMARY:
The purpose of this study is to specifically investigate whether oxytocin and mechanical dilation decreases the rate of cesarean section compared to misoprostol and mechanical dilation for pregnancies at risk of fetal compromise

DETAILED DESCRIPTION:
This is a single center randomized control trial of two arms. Singleton, cephalic, high risk pregnancies will be randomized to either oxytocin with mechanical dilation versus misoprostol with mechanical dilation.

In group A, receiving misoprostol with mechanical dilation, will serve as the control group. Group B, oxytocin with mechanical dilation, will serve as the experimental group. The expected duration of participation begins at induction of labor and concludes at time of delivery.

ELIGIBILITY:
Inclusion Criteria:

* • Age > 18 years old

  * Singleton, or twins with demise of one
  * Cephalic presentation
  * Intact membranes
  * Hypertension (chronic hypertension, gestational hypertension, pre-eclampsia with/without severe features, superimposed preeclampsia with/without severe features, eclampsia, HELLP)
  * Oligohydramnios (AFI< 5cm and/or MVP <2cm)
  * Fetal growth restriction (EFW or AC <10th percentile) with normal or abnormal (elevated, absent, or reversed) Umbilical Artery Dopplers
  * Abnormal antenatal fetal testing (NST, Biophysical profile, decreased fetal movement) prompting induction of labor
  * Suspected placental abruption
  * Poorly controlled pre-gestational diabetes, defined as >50% abnormal glucose values requiring increasing doses of anti-glycemic agents >34 weeks, or requiring delivery
  * Gestational Age > 22 weeks
  * Bishop score < 6

Exclusion Criteria:

* • Prior cesarean delivery

  * Allergy to misoprostol
  * Allergy to oxytocin
  * Allergy to silicone/latex
  * Contraindication to vaginal delivery including placenta or vasa previa, Placenta accreta/increta/percreta, prior uterine rupture, Prior myomectomy entering the uterine cavity and necessitating cesarean delivery, active genital herpes, transverse or oblique fetal lie, umbilical cord prolapse, or HIV viral load >1000 copies/mL

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Rate of Cesarean Delivery | 48 hours
  Total rate of cesarean delivery

SECONDARY OUTCOMES:
The time interval from induction-to-delivey for vaginal deliveries | 48 hours
  Maternal outcome
The number of vaginal births within 24 hours | 24 hours
  Maternal outcome
The number of misoprostol doses received by each participant | 24 hours
  Maternal outcome
The incidence of uterine tachysystole | 24 hours
  Defined as greater than 5 contractions in a ten minute window, averaged over 30 minutes
The rate of each indication for the cesarean delivery | 48 hours
  Indications include non-reassuring fetal hear tones, arrest of dilation, arrest in the 2nd stage of labor etc.
The rate of operative vaginal delivery | 48 hours
  Maternal outcome - includes forceps or vacuum assisted deliveries
The rate of intra-amniotic infection | 48 hours
  Maternal outcome
The rate of postpartum hemorrhage | 24 hours
  Maternal outcome
The rate of Fetal heart rate abnormaliies | 48 hours
  recurrent late decelerations, bradycardia, or prolonged deceleration
The number of patients that received betamethasone for fetal lung maturity and/or magnesium sulfate for fetal neuroprotection | 24 hours
  Maternal outcome
The rate of stillbirth | 48 hours
  Fetal/Neonatal outcome
The total rate of Neonatal Apgar scores less than 7 at 5 minutes | 5 minutes
  Neonatal outcome
The total rate of Neonatal RDS | 96 hours
  Neonatal outcome
The total rate of Neonatal admission to the NICU | 96 hours
  Neonatal outcome
The total rate of neonatal arterial umbilical blood pH < 7.1 | 96 hours
  Neonatal outcome
The rate of neonatal Sepsis | 96 hours
  Neonatal outcome
The rate of Neonatal Death | 96 hours
  Neonatal outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Hafez L, Khanuja K, Mendez-Figueroa H, Al-Kouatly HB, Mascio DD, Chauhan SP, Berghella V. Misoprostol with balloon vs oxytocin with balloon in high-risk pregnancy induction: a randomized controlled trial. Am J Obstet Gynecol MFM. 2023 Dec;5(12):101175. doi: 10.1016/j.ajogmf.2023.101175. Epub 2023 Oct 6. PMID 37806650